CLINICAL TRIAL: NCT01578083
Title: The Neurobiology of Chemotherapy-Induced Cognitive Impairment
Brief Title: Chemotherapy-Induced Cognitive Impairment
Acronym: CICI
Status: Completed | Type: Observational
Sponsor: Jay F. Piccirillo, MD (Other)
Collaborators: Washington University Siteman Cancer Center (Other); Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor-Investigator, Jay F. Piccirillo, MD, Professor, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Other Study IDs: 201203045
Record Dates: First submitted 2012-04-12; First posted 2012-04-16 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2012-04

CONDITIONS: Cognitive Symptoms
Keywords: Chemotherapy; Breast Cancer; Cognitive Impairment; Chemo brain
MeSH Terms: conditions — Neurobehavioral Manifestations; Breast Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cognitive Impairment: With self-report cognitive impairment.
- No Cognitive Impairment: Without self-report cognitive impairment.

SUMMARY:
The investigators overall research hypothesis is that systemic chemotherapy induces structural changes in the white matter of the brain as demonstrated with Diffusion Tensor Imaging (DTI) and functional changes in well-defined cortical neural networks as demonstrated by resting-state functional connectivity MRI (rs-fcMRI). The investigators believe these structural and functional changes are responsible for the cognitive symptoms associated with chemotherapy-induced cognitive impairment (CICI).

The Specific Aim for this study is:

To assess the impact of chemotherapy on structural white matter as defined by DTI and functional cognitive networks as defined by rs-fcMRI by comparing a sample of breast cancer survivors with self-reported CICI to breast cancer survivors without CICI.

Hypothesis: Post-chemotherapy breast cancer patients with self-reported CICI will have abnormal structural connections characterized by DTI-defined disruptions in fractional anisotropy (FA) and mean diffusivity (MD) and abnormal functional connectivity characterized by rs-fcMRI-defined disruptions in cognitive networks when compared to patients without self-reported CICI.

DETAILED DESCRIPTION:
Chemotherapy has been linked to cognitive impairments among breast cancer patients, especially in the domains of executive function (planning and problem solving), attention, learning, and information processing. The etiology of these chemotherapy-associated impairments remains unknown, although recent neuroimaging studies suggest that disruption of white matter integrity may play a role. With continued use of chemotherapy in breast cancer patients, this study's novel use of functional neuroimaging will be significant to better inform practitioners and patients of potential consequences to anticipate and serve as a starting point in the development of therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria (Phase I and II):

  * Participants must be females between 35 and 70 years of age.
  * Participants must have been diagnosed with breast cancer and completed chemotherapy,within the preceding 2 years.
  * Participants must have completed their intended full course of chemotherapy regimen at least 30 days prior to participation.
  * Participants must have been diagnosed with invasive ductal or lobular BrCa Stages I, II, or III (American Joint Committee on Cancer (AJCC) staging manual, 7th edition, 2010).

Inclusion Criteria (Phase II)

* Participants must be able to read, write, and speak English fluently.
* Participants must be able to provide a valid informed consent.
* Participants must have a life expectancy of greater than 6 months at the time they are approached for enrollment.
* Cases - Those who self-report CICI and are in the 75th percentile of scores on the Cognitive Failures Questionnaire (CFQ) and have a global rating of cognition response of "Extremely Affected" or "Strongly Affected"
* Controls - Those whose CFQ scores are in the lowest 25th percentile and who report that their daily life is not affected by cognitive impairment. Controls will be selected so that they are age (within 5 years)-matched to a Case.

Exclusion Criteria:

* • Participants with prior cancer diagnoses of other sites with evidence of active disease within the past year.

  * Participants who have received skull-base radiation treatment within the past year for any reason. Skull-base radiation may contribute to the symptoms of CICI.
  * Participants with active diagnoses of any acute or chronic brain-related neurological conditions that can alter normal brain anatomy or function, including Parkinson's disease, Multiple Sclerosis, Alzheimer's Disease, cerebral infarcts, , history of brain tumor(s), epilepsy, or dementia.
  * Must not have a history of traumatic brain injury (loss of consciousness for > 15 min.)
  * Participants with implanted metal objects not compatible with MRI, electrodes, pacemakers, intracardiac lines, or medication pumps.
  * Participants who weigh over 350 pounds (weight limit on MRI machine).
  * Participants with a history of claustrophobia that will preclude undergoing MRI.
  * Participants with an inability to lie flat for MRI.
  * Any medical condition the PI determines would render the study unsafe or not in the best interest of the patient.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer surviviors from Washington University's Siteman Cancer Center and from community at large.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes in fractional anisotropy (FA) in one or more white matter tracts. | post-chemotherapy. One time measure within one year of final dose of chemotherapy.
  As compared with the controls, the breast cancer patients will show decreased fractional anisotropy (FA) in the frontal and temporal white matter (WM) tracts and.

SECONDARY OUTCOMES:
rs-fcMRI-defined disruptions in cognitive cortical networks | post-chemotherapy: post-chemotherapy. One time measure within one year of final dose of chemotherapy.
  As compared with the controls, the breast cancer patients will show decreased functional integrity of the default mode network [DMN], associated with memory; the dorsal and ventral attention networks [DAN/VAN], involved in attention; and the Cognitive/Control network, involved in executive decision-making
Changes in Mean Diffusivity (MD) in one or more white matter tracks | Post Chemotherapy: post-chemotherapy. One time measure within one year of final dose of chemotherapy.
  As compared with the controls, the breast cancer patients will show increased mean diffusivity (MD) in frontal White Matter (WM).

CONTACTS AND LOCATIONS:
Overall Officials: Jay F. Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Piccirillo JF, Hardin FM, Nicklaus J, Kallogjeri D, Wilson M, Ma CX, Coalson RS, Shimony J, Schlaggar BL. Cognitive impairment after chemotherapy related to atypical network architecture for executive control. Oncology. 2015;88(6):360-8. doi: 10.1159/000370117. Epub 2015 Feb 7. PMID 25678046